CLINICAL TRIAL: NCT04083703
Title: Evaluation of Interbody Cage Insertion in Treatment of Lumbar Disc Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fahd Abdel Sabour Ahmed Mohammed, Resident Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cage in LDP
Record Dates: First submitted 2019-09-02; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Lumbar Disc Herniation
Keywords: Interbody Cage
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Diskectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple lumbar discectomy (Experimental)
  Interventions: Procedure: Interbody cage insertion in lumbar disc prolapse
- Lumbar discectomy with inter vertebral cage (Experimental)
  Interventions: Procedure: Interbody cage insertion in lumbar disc prolapse

INTERVENTIONS:
Procedure: Interbody cage insertion in lumbar disc prolapse — Discectomy alone versus interbody cage insertion in treatment of lumbar disc proapse
  Other Names: Discectomy

SUMMARY:
Comparison between discectomy alone and interbody cage insertion in treatment of lumbar disc prolapse

DETAILED DESCRIPTION:
Discectomy for lumbar disc herniation is one of the most common operation performed worldwide for lumbar-related symptoms. The basic principle of the various techniques is to relieve the nerve root compression induced by the herniation. Over the past 30 years, many technical improvements have decreased operative trauma by reducing incision size, thereby reducing postoperative pain and hospital stay and time off work, while improving clinical outcome. Magnification and illumination systems by microscope and endoscope have been introduced to enable minimally invasive techniques. Lumbar interbody fusion using cages has gained momentum in the recent years after approval of the cages by the FDA (United States Federal Drug Administration) for lumbar interbody insertion. The indications for this procedure remain controversial and include mechanical low back pain, degenerative disc disease, recurrent disc herniation, spondylolisthesis (grade I). In degenerative disc disease or following surgical discectomy, segmental stenosis occurs due to a combination of disc herniation, posterior osteophyte formation, facet overriding and hypertrophy and ligamentum flavum hypertrophy. All these factors combine to compromise the nerve root as it exits through the intervertebral foramen resulting in recurrent radiculopathy. In such cases, Lumbar inter body fusion using cages can open up the intervertebral foramen by maintaining or restoring disc height. On the other hand, there is considerable controversy surrounding the effectiveness of lumbar fusion for the treatment of low back pain. Among the different surgical approaches available, with or without instrumentation, none can be considered the "gold standard". The technique and results of inter body fusion were first reported by Cloward. It did not, however, gain widespread acceptance due to technical difficulties. Insertion of a rectangular bone graft makes it difficult to avoid nerve root trauma resulting in radicular deficit or irritation and dural tears. Non-union or bone graft extrusion were reported as well as bone graft collapse with subsequent segmental stenosis.In the past few years, rigid cages housing autogenous bone have become increasingly popular for the purpose of interbody fusion. Their ease of insertion has decreased the technical difficulties of the earlier Cloward approach and makes the procedure more reproducible. The rigidity of the cages also allows for the preservation of the disc space. Cages are available in a wide variety of shapes and designs, the most common being the cylindrical and rectangular wedge shaped cages.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar disc prolapse one or two levels.
* Patients (age >18 and < 70 years old).
* Patients fit for surgery.

Exclusion Criteria:

* Patients with instability of lumbar spine.
* Patients with degenerative diseases.
* More than two levels
* Patients <18 or >70 years.
* Patients unfit for surgery.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Decrease pain after discectomy and interbody cage insertion. | Base line
  Comparison between preoperative pain with lumbar disc prolapse and posoperative pain improved after Interbody cage insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Abdel Hai Moussa Abdel Latif, prof., Study Director — Assiut University hospital,Neurosurgery department; Ahmed Elsayed Abo Kresha, Assistant Prof., Study Director — Assiut University hospital,Neurosurgery department; Mohamed Elsayed mahmoud, Assistant Prof., Study Director — Assiut University hospital,Neurosurgery department

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/19992171
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/16456311
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3638641/
- See also: Related Info — https://www.europepmc.org/abstract/med/1502649
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/7604342
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/1826546